CLINICAL TRIAL: NCT01521325
Title: A Single-Dose Pilot Study of Radiolabeled Amatuximab (MORAb-009) in Mesothelin Over Expressing Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MORAb-009-006
Record Dates: First submitted 2011-01-07; First posted 2012-01-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Mesothelioma; Pancreatic Cancer; Ovarian Cancer; Non-small Cell Lung Cancer
MeSH Terms: conditions — Mesothelioma; Pancreatic Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — amatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amatuximab infusion (Experimental): Subjects will receive one infusion of radiolabeled amatuximab.
  Interventions: Drug: Amatuximab

INTERVENTIONS:
Drug: Amatuximab — Subjects will receive one infusion of radiolabeled amatuximab.
  Other Names: MORAb-009; MORAB-009-006

SUMMARY:
This research is being conducted to determine the biodistribution of radiolabeled amatuximab in tumor and non-tumor tissues in subjects with mesothelin over expressing cancer including mesothelioma, pancreatic, ovarian or non small cell lung cancer.

DETAILED DESCRIPTION:
The primary objective is to determine the biodistribution of radiolabeled amatuximab in tumor and nontumor tissues in subjects with mesothelin over-expressing cancers including mesothelioma, pancreatic, ovarian, and non small cell lung cancer. This is a single-center, single-dose, open-label, pilot study of amatuximab in approximately 20 subjects with mesothelin expressing tumors. 111Indium-radiolabeled amatuximab (5 mCi) will be administered. Serial SPECT imaging (at 3 specific time points up to 196 hours after cold infusion) will be performed to determine binding to tumor and nontumor tissue. Subjects will be observed closely for safety and possible development of anti-amatuximab antibodies. Pharmacokinetics of radiolabeled antibody will be determined with imaging over time.

ELIGIBILITY:
Inclusion Criteria:

* Female and Male subjects > or = 18 years of age
* Histologically confirmed mesothelin-expressing cancer
* Measurable disease that has progressed through prior therapy and that includes a non-hepatic lesion for imaging that is > or = 1.5cm, as defined by RECIST v1.1 and disease location, at discretion of the physician, or evaluable by clinical symptoms supported by biomarker, radiological or pathological studies conducted within 4 weeks prior to study entry

Exclusion Criteria:

* Known allergy or hypersensitivity to monoclonal antibodies
* Known to develop HACA
* Prior treatment with amatuximab
* Prior treatment with SS1 (dsFv)PE38 (ss1P)
* Prior treatment with another test article within previous 30 days
* Known brain metastasis
* Known prosthetic devices that would prohibit imaging ow lesion of interest due to radiographic artifact
* Chemotherapy, biological therapy, radiation therapy or immunotherapy within 3 weeks prior to dosing with amatuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Primary Objective: determine biodistribution of radiolabeled amatuximab in tumor and nontumor tissue | 1 year
  To determine the biodistribution of radiolabeled amatuximab in tumor and nontumor tissue in subjects with mesothelin over expressing cancer including mesothelioma, pancreatic, ovarian or nonsmall cell lung cancer by performing SPECT imaging to determine binding to tumor and non-tumor tissue.

SECONDARY OUTCOMES:
Secondary objectives: determine the safety of a single IV of Indium-CHX-A amatuximab | 1 year
  To determine the safety of a single IV of Indium-CHX-A amatuximab by collecting safety data during/ after the infusions as well as obtain any potential drug-related AEs 30 days post infusion
Pharmacokinetic and serum levels | 1 year
  To determine the PK parameters of the Indium-CHX-A amatuximab with imaging, and serum levels collected over time
uptake of Indium-CHX-A amatuximab | 1 year
  To explore the uptake of Indium-CHX-A amatuximab with mesothelin tumor expression as determined by ICH
occurrence of HACA | 1 year
  To tabulate the occurrence of HACA which will be measured through serum samples collected over time
correlate shed serum mesothelin to imaging | 1 year
  To correlate shed serum mesothelin to imaging obtained after antibody administration.

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, MD, Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Cacner Institue, Bethesda, Maryland, United States